CLINICAL TRIAL: NCT04126590
Title: Phase I Clinical Study of Safety，Tolerability， Pharmacokinetics and Pharmacodynamics of Recombinant Humanized Cytotoxic T Lymphocyte Antigen 4 Single Domain Antibody Fc Fusion Protein Injection in Subjects With Advanced Solid Tumors
Brief Title: Phase I Study of KN044 in Locally Advanced/Metastatic Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun Intellicrown Pharmaceutical Co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KN0440101a
Record Dates: First submitted 2019-10-10; First posted 2019-10-15 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Advanced Solid Tumors
Keywords: Adverse Event; Anti-Drug Antibodies; Complete Response
MeSH Terms: conditions — Pathologic Complete Response

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- KN044 0.03 mg/kg dose group (Experimental): KN044 0.03 mg/kg dose group,once every 3 weeks，a total of four cycles
  Interventions: Biological: KN044
- KN044 0.1 mg/kg dose group (Experimental): KN044 0.1 mg/kg dose group,once every 3 weeks，a total of four cycles
  Interventions: Biological: KN044
- KN044 0.3mg/kg dose group (Experimental): KN044 0.3mg/kg dose group,once every 3 weeks，a total of four cycles
  Interventions: Biological: KN044
- KN044 1 mg/kg dose group (Experimental): KN044 1 mg/kg dose group,once every 3 weeks，a total of four cycles
  Interventions: Biological: KN044
- KN044 3 mg/kg dose group (Experimental): KN044 3 mg/kg dose group,once every 3 weeks，a total of four cycles
  Interventions: Biological: KN044
- KN044 6mg/kg dose group (Experimental): KN044 6mg/kg dose group,once every 3 weeks，a total of four cycles
  Interventions: Biological: KN044
- KN044 10mg/kg dose group (Experimental): KN044 10mg/kg dose group,once every 3 weeks，a total of four cycles
  Interventions: Biological: KN044

INTERVENTIONS:
Biological: KN044 — The modified phase I "3 + 3" study design was used in dose escalation from low dose to high dose to determine the MTD.Sequential assignment of Patient cohorts to one of five dose levels of KN044: 0.03mg/kg,0.3 mg/kg,1 mg/kg,3 mg/kg,6 mg/kg,10 mg/kg.

SUMMARY:
This is an open-label, multicenter, dose-escalation phase I study to assess the safety, tolerability and preliminary efficacy of KN044 in participants with all advanced solid tumors who are not able to have current standard anti-tumor therapies. The purpose of this study is to determine the maximum tolerated dose (MTD) , to characterise the safety, pharmacokinetics (PK), immunogenicity, pharmacodynamics (PD) and anti-tumor activity of KN044 as a single agent in adult participants with advanced solid tumors.

DETAILED DESCRIPTION:
This study will involve patients and follow the standard "3 + 3"design. KN044 will be antimedical intravenously over 30 minutes with planned doses of 0.03, 0.1, 0.3, 1, 3, 6,10 mg/kg Once every 3 weeks for first 4 doses, then every 3, or 6, or 12 weeks for up to 1 year if no intolerable toxicities occur and per agreement with investigator antimedical monitor based on emerging data.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects can understand informed consent, voluntarily participate and sign informed consent.
2. Tumor subject type Clinical diagnosis of advanced malignant tumors. Patients diagnosed by pathology and/or cytology; malignant melanoma, patients with advanced renal cell carcinoma, colorectal cancer, lung cancer, breast cancer, prostate cancer, etc. are preferred; the inclusion of melanoma is pathological and / or cytologically undiagnosed unresectable patients with stage 3b/3c or stage 4 (M1a / M1b) melanoma, in which patients with stage IV M1b have to meet the following requirements: no more than 5; the longest path of a single lesion must not exceed 20 mm; the sum of the longest diameters of the cumulative lesions must not exceed 50 mm.
3. Subjects with locally advanced (non-resectable) and / or metastatic solid tumor that has progressed after standard therapies or no standard therapy exists.
4. Previous anti-tumor therapy (including endocrine chemoradiotherapy/radiotherapy, targeted therapy) ended more than 4 weeks and has been restored to baseline or ≤ grade 1 from previous adverse events following [Common Criteria for Assessment of Adverse Events (CTCAE) version 5.0] (except for patients with hair loss).
5. 18-75 years of age, male or female; 10)Eastern Cooperative Oncology Group score 0 or 2; Life expectancy ≥ 3 months.
6. Previous major surgery ≥1 month ago.
7. Must have adequate organ function, prior to start of KN044, including the following:

   1. white blood cell count ≥ 3.0 × 109 / L;
   2. absolute neutrophil count (ANC) ≥ 1.5 ×109/L;
   3. platelet count ≥ 100 × 109/L;
   4. hemoglobin ≥ 9 g/dL
   5. serum albumin ≥ 2.5 g / dL;
   6. Hepatic: total bilirubin ≤ 1.5 times the upper limit of normal (ULN); aspartate transaminase (AST) and/or alanine aminotransferase (ALT) ≤ 2.5× ULN (≤5 × ULN if with liver involvement)
   7. Renal: Serum creatinine ≤ 1.5×ULN or 24-hour Estimated clearance≥50 mL / min (Cockcroft and Gault formula);
   8. Coagulation tests International standardization ratio (INR) ≤ 1.5, prothrombin time (PT), activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN
8. Normal left ventricular ejection fraction (LVEF) ≥50% measured by multigated radionuclide angiography or Echocardiography.
9. Female patient with fertility or male patient whose partner has fertility should use one or more contraceptive methods for contraception within at least eight months from the screening period to five half-lives after the last treatment. These measures include, but are not limited to, oral or implantable injections of hormonal contraceptives; intrauterine birth control ring or placement of hormone-releasing intrauterine device); or use of barrier methods such as condoms or septum and spermicide products.
10. According to ResponseEvaluationCriteriainSolid Tumors Version1.1, the subject should have an assessable lesion (target lesion or non-target lesion)
11. grade ≤ 2 peripheral neuropathy can be enrolled

Exclusion Criteria:

1. At the discretion of the investigator, there are both serious medical conditions that may harm the safety of the subject or affect the subject's completion of the study, including but not limited to: severe heart disease, cerebrovascular disease, uncontrolled diabetes, Insulin dependent diabetes, serious infection;Thyroid disease
2. Accepted any other anti-tumor drug therapies, or other immunological anti-tumor treatments, including but not limited to PD-1/L1 inhibitors before the first KN044 dosing.
3. Pregnant or nursing females
4. Severe or uncontrolled cardiac disease requiring treatment, congestive heart failure New York Heart Association III or IV, unstable angina pectoris even if medically controlled, history of myocardial infarction during the last 6 months, ECG QT interval（fridericia)> 450msec, serious arrhythmias requiring medication (with exception of atrial fibrillation or paroxysmal supraventricular tachycardia)；Hypertension (defined as sustained systolic blood pressure> 150 mm Hg and / or post-diastolic blood pressure with antihypertensive drugs> 100 mm Hg;
5. suffering from mental disorders, infectious diseases, and skin diseases that are difficult to control;
6. Known active hepatitis B or C or known infection with HIV .
7. History of life-threatening hypersensitivity, or known to be allergic to protein drugs or recombinant proteins or any ingredients in KN044 drug formulation
8. Known severe bleeding factors that can affect venous blood sampling;
9. Acute or chronic uncontrolled renal disease, pancreatitis or liver disease (per investigator assessment).
10. Subjects with active autoimmune disease or a documented medical history of autoimmune disease or symptoms that require systemic use of steroid and/or immunosuppressant. Exceptions are subjects with vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus or hypothyroidism which can be managed by replacement therapy.
11. Use of more than 15 mg of prednisone or equivalent dose of steroids per day within 3 months of administration.
12. Electrocardiogram QT interval (fridericia) > 450 msec and severe arrhythmia requiring medication (except for atrial fibrillation or paroxysmal supraventricular tachycardia);
13. Uncontrolled primary central nervous system tumors or central nervous system metastasis; based on screening brain magnetic resonance imaging (MRI), patients who have one of the following may not be excluded:

    1. No evidence of brain metastases or has to be clinically stable for at least 4 weeks
    2. Untreated brain metastases not needing immediate local therapy
14. Live vaccines are banned 30 days prior to enrollment and during clinical studies. Inactive vaccines are allowed during the study;
15. Within 30 days prior to screening, the patient has undergone any other experimental drug therapy or has participated in another interventional clinical trial;
16. The study may not be completed for other reasons or the Investigators believes that it should not be included;
17. Peripheral neuropathy >Grade 2.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-01-09 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity for The maximum tolerated dose | up to 6 weeks
  Dose-limiting toxicity observation period 6 weeks after the first dose
KN044 of adverse event | through study completion, an average of 210 days
  the adverse events are recorded according to the actual occurrence
KN044 of abnormalities of physical findings and laboratory tests, | through study completion, an average of 210 days
  The data of the clinical research center is collected and analyzed according to the time point of the test flow chart

SECONDARY OUTCOMES:
PK parameters: Area under curve (AUC) | an average of 126 days
  According to the test schedule, the blood volume of each subject's PK was analyzed and PK analysis was performed.
PK parameters: Cmax | an average of 126 days
  According to the test schedule, the blood volume of each subject's PK was analyzed and PK analysis was performed.
PK parameters: Clearance rate (CL) | an average of 126 days
  According to the test schedule, the blood volume of each subject's PK was analyzed and PK analysis was performed.
PK parameters: t1/2 | an average of 126 days
  According to the test schedule, the blood volume of each subject's PK was analyzed and PK analysis was performed.
PK parameters: Vss | an average of 126 days
  According to the test schedule, the blood volume of each subject's PK was analyzed and PK analysis was performed.
PK parameters: dose proportionality | an average of 126 days
  According to the test schedule, the blood volume of each subject's PK was analyzed and PK analysis was performed.
Incidence of the positive anti-drug antibodies and titers of anti-drug antibodies | an average of 147 days
  According to the test schedule, the blood volume of each subject's anti-drug antibodies was analyzed and anti-drug antibodies analysis was performed.
Anti-tumor activity as measured by ResponseEvaluationCriteriainSolidTumors Version1.1(RESISTv1.1) | During the treatment period , the tumor was evaluated every 6 weeks, then every 9 weeks.
  Evaluation of tumor response according to RESISTv1.1 criteria, complete relief（CR), Partial relief(PR), Stable disease(SD), PD、ORR[CR＋PR]）、Disease control rate(DCR[CR＋PR＋SD]）、PFS、DOR

CONTACTS AND LOCATIONS:
Overall Officials: chunmei Bai, Principal Investigator — Peking Union Medical College Hospital; Rui Chen, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No